CLINICAL TRIAL: NCT01093456
Title: Diurnal Variation of Mineral Metabolism and Protein Fermentation Metabolites in Peritoneal Dialysis Patients and Healthy Volunteers
Brief Title: Diurnal Variation of Uremic Solutes in Peritoneal Dialysis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML6275
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Kidney Disease
Keywords: diurnal variation; peritoneal dialysis; uremic retention solutes; phosphorous; indoxyl sulfate; p-cresol sulfate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood, serum, urine and dialysate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- chronic kidney disease: ESKD patients treated with peritoneal dialysis
- Healthy volunteers: healthy volunteers, aged 18 years and above

SUMMARY:
Study on the daytime variation of uremic retention solutes and markers of bone-mineral metabolism in patients with end-stage kidney disease treated with peritoneal dialysis

DETAILED DESCRIPTION:
Many epidemiological studies have pointed to the association between serum parameters of phosphate metabolism (phosphate, FGF23) and microbiotic protein fermentation (p-cresyl sulphate [PCS], indoxyl sulphate [IS]) on the one hand and increased risk of all-cause and cardiovascular death on the other hand.

Hypothesis: Due to failing feed-back mechanisms, diurnal variation of serum concentrations of serum phosphate and fermentation metabolites will be more pronounced in dialysis patients, especially in those with negligible residual kidney function.

Clinical studies assessing this issue are scarce to non-existing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Normal dietary habits

Exclusion Criteria:

* Treatment with systemic antibiotics within one month Major abdominal surgery Drugs known to affect gastrointestinal physiology (acid secretion inhibitors, prokinetics, laxatives, probiotics, prebiotics,..)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Peritoneal dialysis patients Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the diurnal variation of serum concentrations of phosphate and protein fermentation metabolites in healthy volunteers as compared to dialysis patients. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Evenepoel, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospital, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No